CLINICAL TRIAL: NCT06284421
Title: Use of a Durometer to Measure Uterine Tone in Cesarean Delivery
Brief Title: Durometer for Measuring Uterine Tone
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB23-1068
Record Dates: First submitted 2024-02-13; First posted 2024-02-29 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Uterine Tone Disorders; Cesarean Section Complications

STUDY DESIGN:
Intervention Model Description: To determine the feasibility of using a portable, digital Shore OO durometer to measure uterine tone during elective cesarean delivery. We hypothesize that this durometer will be easy to use by operating obstetricians for the measurement of uterine tone during cesarean delivery. Also we hope to be to correlate the hardness of uterine tone, as measured by the Shore OO durometer, with a 0-10 score on the uterine tone score and the administration of extra uterotonic drugs for uterine atony. [NB- the administration of extra uterotonic drugs is dependent on the clinical decision made by the obstetrician in agreement with the anesthesiologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Durometer (Experimental): This is a single-arm trial in which a Shore durometer will be used to measure the hardness of the uterus after placental delivery during cesarean section.
  Interventions: Device: Shore durometer

INTERVENTIONS:
Device: Shore durometer — The durometer will be held on the exterior of the lower uterine segment and fundus to measure the hardness reading at each location.

SUMMARY:
This study will evaluate the use of a durometer to measure uterine tone in parturients undergoing cesarean delivery.

DETAILED DESCRIPTION:
The most accurate and precise measure of uterine tone is unknown. The most commonly described in vivo method in the literature is a qualitative numeric scoring scale from 0-10. The 0-10 uterine tone score has demonstrated good and excellent inter-rater reliability between 1 and 2 raters respectively, and good inter-rater agreement. Recent data suggests that the 0-10 uterine tone score is well-correlated with clinical assessments of uterine tone.

A handful of studies have used a quantitative "hardness meter", including a Shore durometer, to describe uterine tone in vivo, with promising results. The instrument has not yet been validated in cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Non-emergent (scheduled) cesarean delivery at University of Chicago Family Birth Center
* Patients ages 18-50

Exclusion Criteria:

* Patients undergoing unscheduled (intrapartum) cesarean delivery
* Ages <18 or >50 years old
* Intrapartum cesarean hysterectomy
* Inability to provide independent, informed consent due to impairment or intellectual disability
* Non-English speaking patients

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
feasibility of a durometer | within 10 minutes after placental delivery
  The primary outcome will be the ability to obtain reliable readings of the 'hardness' of the uterus during a cesarean delivery.

SECONDARY OUTCOMES:
durometer reading | 0 minutes after placental delivery
  average durometer reading at lower uterine segment and fundus
durometer reading | 3 minutes after placental delivery
  average durometer reading at lower uterine segment and fundus
durometer reading | 10 minutes after placental delivery
  average durometer reading at lower uterine segment and fundus
correlation of durometer reading with a 0-10 uterine tone rating score (0= "no tone"; 10= "excellent tone") | 0 minutes after placental delivery
  correlation of 2 measures
correlation of durometer reading with a 0-10 uterine tone rating score (0= "no tone"; 10= "excellent tone") | 3 minutes after placental delivery
  correlation of 2 measures
correlation of durometer reading with a 0-10 uterine tone rating score (0= "no tone"; 10= "excellent tone") | 10 minutes after placental delivery
  correlation of 2 measures

CONTACTS AND LOCATIONS:
Overall Officials: Naida Cole, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No